CLINICAL TRIAL: NCT03435250
Title: A Phase 1 Study of AG-270 in the Treatment of Subjects With Advanced Solid Tumors or Lymphoma With Homozygous Deletion of MTAP
Brief Title: Study of AG-270 in Participants With Advanced Solid Tumors or Lymphoma With MTAP Loss
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic reasons
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG270-C-001
Record Dates: First submitted 2018-02-01; First posted 2018-02-19 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumors; Lymphoma
Keywords: MTAP; MTAP deletion; CDKN2A deletion; MAT2A inhibitor; Advanced solid tumors; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Docetaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AG-270 (Experimental): AG-270 will be administered on Days 1 to 28 of each 28-day cycle. Treatment will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: AG-270
- AG-270/docetaxel (Experimental): AG-270 will be administered daily, starting 1 week prior to docetaxel infusion. Starting on Cycle 1 Day 1, docetaxel (by intravenous infusion [IV]) will be administered once during each 21-day cycle. Treatment with AG-270 and docetaxel will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: AG-270; Drug: docetaxel
- AG-270/nab-paclitaxel/gemcitabine (Experimental): AG-270 will be administered daily, starting 1 week prior to nab-paclitaxel and gemcitabine infusion. Starting on Cycle 1 Day 1, nab-paclitaxel and gemcitabine IV will be administered on Days 1,8, and 15 during each 28-day cycle. Treatment with AG-270, nab-paclitaxel, and gemcitabine will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: AG-270; Drug: nab-paclitaxel; Drug: gemcitabine

INTERVENTIONS:
Drug: AG-270 — AG-270, orally, once or twice daily, on Days 1 through 28 of each 28-day cycle, until disease progression or unacceptable toxicity.
  Other Names: MAT2A inhibitor
  Arms: AG-270
Drug: AG-270 — AG-270, orally, once or twice daily, for 1 week prior to the first dose of docetaxel. Thereafter, AG-270 continues to be given daily, on Days 1 through 21 of each 21-day cycle, until disease progression or unacceptable toxicity.
  Other Names: MAT2A inhibitor
  Arms: AG-270/docetaxel
Drug: AG-270 — AG-270, orally, once or twice daily for 1 week prior to the first doses of nab-paclitaxel and gemcitabine. Thereafter, AG-270 continues to be given daily on Days 1 through 28 of each 28-day cycle, until disease progression or unacceptable toxicity.
  Other Names: MAT2A inhibitor
  Arms: AG-270/nab-paclitaxel/gemcitabine
Drug: docetaxel — Docetaxel, IV, once during each 21-day cycle, until disease progression or unacceptable toxicity.
  Other Names: Taxotere®
  Arms: AG-270/docetaxel
Drug: nab-paclitaxel — Nab-paclitaxel, IV, on Days 1, 8, and 15 of each 28-day cycle, until disease progression or unacceptable toxicity.
  Other Names: Abraxane®
  Arms: AG-270/nab-paclitaxel/gemcitabine
Drug: gemcitabine — Gemcitabine, IV, on Days 1, 8, and 15 of each 28-day cycle, until disease progression or unacceptable toxicity.
  Other Names: Gemzar®
  Arms: AG-270/nab-paclitaxel/gemcitabine

SUMMARY:
This study will evaluate the safety, pharmacokinetics, pharmacodynamics, and clinical activity of AG-270 in participants with advanced solid tumors or lymphoma with homozygous MTAP deletion.

DETAILED DESCRIPTION:
The purpose of this Phase 1, multicenter, open-label study is to determine the maximum tolerated dose (MTD) of AG-270, administered as a single agent or in combination with taxane-based chemotherapy, and to characterize its dose-limiting toxicities (DLTs) when given daily by mouth to participants with advanced solid tumors or lymphoma with homozygous deletion of methylthioadenosine phosphorylase (MTAP).

In each arm of the study, successive cohorts of participants will receive increasing oral doses of AG-270 to determine the MTD, the dose with maximum pharmacologic activity or the maximum feasible dose, as a single agent and in combination with taxane-based chemotherapy. In the subsequent dose-expansion parts of the study, additional participants in each treatment arm will be treated at the MTD (or one of the described alternative doses) to further characterize that dose's safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD), and to detect preliminary evidence of anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

AG-270 Monotherapy

1. Be ≥18 years of age;
2. Have a histologically confirmed diagnosis of an advanced solid tumor or lymphoma that has progressed in spite of at least one prior line of treatment, and for which additional effective standard therapy is not available. For this study, effective standard therapy is defined as treatment that has been shown to be curative and/or to prolong survival. In addition, participants who are considered to not be candidates for standard therapy or who decline standard therapy are eligible for this study; in such cases, documentation of the reason for omitting or declining a standard therapy is required;
3. Have evidence of homozygous loss of cyclin-dependent kinase inhibitor 2A (CDKN2A) and/or MTAP in the participant's tumor tissue;
4. Have disease that can be clinically evaluated for improvement or progression. In the dose-expansion phase of the study arm, participants must have disease that is measurable, as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria for solid tumors (Eisenhauer et al, 2009) or the Lugano criteria for lymphoma (Cheson et al, 2014);
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤2;
6. Have a hemoglobin ≥9.0 grams per deciliter (g/dL) without red blood cell transfusion for ≥1 month;
7. Have an absolute neutrophil count (ANC) ≥1.0 × 10^9/liter (L);
8. Have a platelet count ≥75 × 10^9/L;
9. Have a serum total bilirubin ≤1.5 × upper limit of normal (ULN);
10. Have an alanine aminotransferase (ALT) ≤3.0 × ULN. (Note: There are no specific requirements for aspartate aminotransferase (AST) or Alkaline phosphatase [ALP]);
11. Have a serum creatinine ≤1.5 × ULN;
12. Be fully recovered from major surgery and from the acute toxic effects of prior chemotherapy and radiotherapy. Residual chronic toxicities of prior therapy ≤Grade 2 (eg, peripheral neuropathy, residual alopecia) are allowed;
13. Female participants who are pre-menopausal or have experienced menopause for less than 2 years and who have not undergone a hysterectomy, bilateral oophorectomy, or tubal occlusion must have a negative serum pregnancy test during screening and a serum or urine pregnancy test must be re-confirmed as negative no more than 72 hours before starting AG-270. Females of reproductive potential as well as fertile men with partners who are female of reproductive potential must agree to abstain from sexual intercourse or to use 2 effective forms of contraception (including at least 1 barrier form) from the time of giving informed consent, during the study, and for 6 months (for females) and for 3 months (for males) following the last dose of AG-270. Effective forms of contraception are defined as hormonal oral contraceptives, injectables, patches, intrauterine devices, double-barrier methods (eg, synthetic condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), or male partner sterilization;
14. Able to understand and has provided written informed consent. A legally authorized representative may consent on behalf of a participant who is otherwise unable to provide informed consent, if acceptable to and approved by the site and/or site's Institutional Review Board (IRB)/Independent Ethics Committee (IEC).

AG-270 in Combination with Docetaxel

1. a. Be ≥18 years of age;
2. a. Have histologically confirmed diagnosis of non-small cell lung cancer (NSCLC) that has been treated with no more than 2 prior lines of cytotoxic chemotherapy in the setting of metastatic (Stage 4) disease. Three prior lines of cytotoxic chemotherapy for metastatic disease are allowed if one of the 3 lines was a maintenance treatment. Participants with solid tumors other than NSCLC for which docetaxel is indicated are eligible for the dose-escalation arm, but they also must have received no more than 2 prior lines of cytotoxic chemotherapy in the setting of metastatic disease; For both participants with NSCLC and participants with other malignancies prior treatment with taxanes is permitted, but prior treatment with docetaxel is not allowed. There is no limitation on the number of non-cytotoxic therapies that a participant with NSCLC or with another malignancy may have received;
3. a. Have evidence of homozygous loss of CDKN2A and/or MTAP in the participant's tumor tissue. In the dose expansion phase of the combination, participants must have homozygous MTAP deletion;
4. a. Have disease that can be clinically evaluated for improvement or progression. In the dose-expansion phase of this study arm, participants must have disease that is measurable, as defined by the RECIST Version 1.1 criteria for solid tumors (Eisenhauer et al, 2009);
5. a. Have an ECOG PS of ≤1;
6. a. Have a hemoglobin ≥9.0 g/dL without red blood cell transfusion for ≥1 month;
7. a. Have an ANC ≥1.5 × 10^9/L;
8. a. Have a platelet count ≥100 × 10^9/L;
9. a. Have a serum total bilirubin ≤1.5 × ULN;
10. a. Have an ALT ≤3.0 × ULN. If ALP is >2.5 × ULN and the increase in ALP cannot be attributed to bone metastases or other bone disease then the participant must have ALT and AST values that are both <1.0 × ULN; this requirement conforms with the current label for Taxotere®;
11. a. Have a serum creatinine ≤1.5 × ULN;
12. a. Meet any criteria necessary for the safe and proper use of docetaxel;
13. a. Be fully recovered from major surgery and from the acute toxic effects of prior chemotherapy and radiotherapy. Residual chronic toxicities of prior therapy ≤ Grade 2 (eg, peripheral neuropathy, residual alopecia) are allowed;
14. a. Female participants who are pre-menopausal or have experienced menopause for less than 2 years and who have not undergone a hysterectomy, bilateral oophorectomy, or tubal occlusion must have a negative serum pregnancy test during Screening and a serum or urine pregnancy test must be re-confirmed as negative no more than 72 hours before starting AG-270. Females of reproductive potential as well as fertile men with partners who are female of reproductive potential must agree to abstain from sexual intercourse or to use 2 effective forms of contraception (including at least 1 barrier form) from the time of giving informed consent, during the study, and for 6 months (for females) and for 3 months (for males) following the last dose of AG-270. Effective forms of contraception are defined as hormonal oral contraceptives, injectables, patches, intrauterine devices, double-barrier methods (eg, synthetic condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), or male partner sterilization;
15. a. Able to understand and has provided written informed consent. A legally authorized representative may consent on behalf of a participant who is otherwise unable to provide informed consent, if acceptable to and approved by the site and/or site's IRB/IEC.

AG-270 in Combination with nab-Paclitaxel and Gemcitabine

1. b. Be ≥18 years of age;
2. b. Have locally advanced or metastatic pancreatic ductal adenocarcinoma characterized by CDKN2A deletion and/or MTAP deletion;
3. b. Have evidence of homozygous loss of CDKN2A and/or MTAP in the participant's tumor tissue. In the dose expansion phase of the combination, participants must have homozygous MTAP deletion;
4. b. Have received no more than 1 previous line of cytotoxic chemotherapy for advanced or metastatic disease. Participants may have been treated with cytotoxic chemotherapy in the adjuvant setting if the final dose of such adjuvant treatment was given at least 6 months before administration of the first doses of AG-270, nab-paclitaxel, and gemcitabine; treatment with cytotoxic chemotherapy in the adjuvant setting will not be counted in the lines of previous cytotoxic chemotherapy for advanced or metastatic disease. There is no limitation on the number of non-cytotoxic therapies that a participant may have received;
5. b. Have an ECOG PS of ≤1;
6. b. Have a hemoglobin ≥9.0 g/dL without red blood cell transfusion for ≥1 month;
7. b. Have an ANC ≥1.5 × 10^9/L;
8. b. Have a platelet count ≥100 × 10^9/L;
9. b. Have a serum total bilirubin ≤1.5 × ULN;
10. b. Have an ALT ≤3.0 × ULN. (Note: There are no specific requirements for AST or ALP.);
11. b. Have a serum creatinine ≤1.5 × ULN;
12. b. Meet any criteria necessary for the safe and proper use of nab-paclitaxel and gemcitabine;
13. b. Be fully recovered from major surgery and from the acute toxic effects of prior chemotherapy and radiotherapy. Residual chronic toxicities of prior therapy ≤ Grade 2 (eg, peripheral neuropathy, residual alopecia) are allowed;
14. b. Female participants who are pre-menopausal or have experienced menopause for less than 2 years and who have not undergone a hysterectomy, bilateral oophorectomy, or tubal occlusion must have a negative serum pregnancy test during Screening and a serum or urine pregnancy test must be re-confirmed as negative no more than 72 hours before starting AG-270. Females of reproductive potential as well as fertile men with partners who are female of reproductive potential must agree to abstain from sexual intercourse or to use 2 effective forms of contraception (including at least 1 barrier form) from the time of giving informed consent, during the study, and for 6 months (for females) and for 3 months (for males) following the last dose of AG-270. Effective forms of contraception are defined as hormonal oral contraceptives, injectables, patches, intrauterine devices, double-barrier methods (eg, synthetic condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), or male partner sterilization;
15. b. Able to understand and has provided written informed consent. A legally authorized representative may consent on behalf of a participant who is otherwise unable to provide informed consent, if acceptable to and approved by the site and/or site's IRB/IEC.

Exclusion Criteria (All Treatment Arms):

1. Have a primary central nervous system (CNS) malignancy (eg, glioblastoma multiforme [GBM]);
2. Have metastasis to the CNS that is symptomatic and/or requires therapy with corticosteroids or anti-convulsant medication. However, participants who have completed treatment (radiation therapy) for CNS metastases and do not require continued treatment with corticosteroids or anti-convulsants may be enrolled in this study;
3. Have a history of Gilbert's syndrome;
4. Have a degenerative retinal disease. Retinal diseases that require a participant's exclusion include: glaucoma (with the exception of narrow angle glaucoma), hereditary retinal diseases such as retinitis pigmentosa; retinal arterial occlusive disease; and retinal disease with advanced scarring, to include age-related macular degeneration and myopic degeneration with geographic atrophy;
5. Have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of AG-270, including any unresolved nausea, vomiting, or diarrhea that is National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade >1;
6. Have had significant active cardiac disease within 6 months prior to the start of study treatment, including any of the following:

   1. New York Heart Association (NYHA) class III or IV congestive heart failure;
   2. Acute myocardial infarction or angina pectoris;
   3. Stroke;
   4. Uncontrolled cardiac arrhythmia (participants with rate-controlled atrial fibrillation are not excluded).
7. Have a heart-rate corrected QT interval using Fridericia's method (QTcF) >470 milliseconds (msec);
8. Have any other concurrent severe and/or uncontrolled concomitant medical condition that could compromise participation in the study (eg, clinically significant pulmonary disease, clinically significant neurological disorder, active or uncontrolled infection);
9. Have received systemic anti-cancer treatment or radiotherapy less than 2 weeks before the first dose of AG-270. Participants with castration-resistant prostate cancer may continue therapy with a luteinizing hormone releasing hormone (LHRH) agonist while participating in this study. Continuation of supportive therapy with bisphosphonates or denosumab is also allowed, regardless of the underlying malignancy;
10. Have received radioimmunotherapy (eg, 131I-tositumomab, 90Y-ibritumomab tiuxetan) less than 6 weeks before the first dose of AG-270;
11. Have received treatment with a therapeutic antibody less than 4 weeks before the first dose of AG-270. A minimum 2-week period between the last treatment with a therapeutic antibody and the first dose of AG-270 may be permitted in participants with rapidly progressive or aggressive subtypes of lymphoma following discussion with the medical monitor;
12. Have received treatment with an investigational small molecule less than 2 weeks before the first dose of AG-270. In addition, the first dose of AG-270 should not occur before a period greater than or equal to 5 half-lives of the investigational small molecule has elapsed;
13. Require continued treatment with a medication that is known to be a strong inhibitor of cytochrome P450 (CYP)3A enzymes. (Treatment with moderate or weak CYP enzyme inhibitors is allowed.);
14. Require continued treatment with a medication that is known to be a strong inducer of CYP3A;
15. Require continued treatment with a medication that is known to be a strong inhibitor of CYP2C8;
16. Require continued treatment with a medication that is a sensitive CYP2C9 substrate with a narrow therapeutic index;
17. Require continued treatment with medications that are known to carry a risk of torsades de pointes;
18. Are pregnant or breastfeeding;
19. Have any other medical or psychological condition deemed by the Investigator to likely interfere with the participant's ability to give informed consent or participate in the study;
20. Are unable to take no food or liquids other than water for 2 hours before and 2 hours after each dose of AG-270.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-03-04 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with DLTs Associated with AG-270 Administration During the First Cycle (First 28 Days) of Treatment | Up to 28 days, on average
Percentage of Participants with DLTs Associated with the Combination of AG-270 and Docetaxel Administration During the First Cycle (First 28 Days) of Treatment | Up to 28 days, on average
Percentage of Participants with DLTs Associated with the Combination of AG-270, nab-paclitaxel, and Gemcitabine Administration During the First Cycle (First 28 Days) of Treatment | Up to 28 days, on average

SECONDARY OUTCOMES:
Percentage of Participants with Treatment-related Adverse Events and Serious Adverse Events | Up to 30 weeks, on average
Changes in Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) Score | Up to 30 weeks, on average
Area under the Concentration-versus-time Curve (AUC) from 0 to Time of Last Measurable Concentration (AUC0-t) of AG-270 | At multiple time points up to 30 weeks, on average
AUC from 0 to Infinity (AUC0-∞) of AG-270 | At multiple time points up to 30 weeks, on average
AUC over One Dosing Interval at Steady State (AUCtau,ss) of AG-270 | At multiple time points up to 30 weeks, on average
Time to Maximum Concentration (Tmax) of AG-270 | At multiple time points up to 30 weeks, on average
Maximum Concentration (Cmax) of AG-270 | At multiple time points up to 30 weeks, on average
Trough Concentration (Ctrough) of AG-270 | At multiple time points up to 30 weeks, on average
Half-life (t1/2) of AG-270 | At multiple time points up to 30 weeks, on average
Apparent Volume of Distribution (Vd/F) of AG-270 | At multiple time points up to 30 weeks, on average
Apparent Clearance (CL/F) of AG-270 | At multiple time points up to 30 weeks, on average
Change from Baseline in Circulating Concentration of S-adenosylmethionine (SAM) | Up to 30 weeks, on average
Change from Baseline in Circulating Concentration of Methionine | Up to 30 weeks, on average
Clinical Activity of AG-270 in Solid Tumors as Assessed by RECIST V1.1 | Up to 30 weeks, on average
Clinical Activity of AG-270 in Lymphoma as Assessed by Lugano Criteria | Up to 30 weeks, on average
Duration of Response (DOR) | Up to 30 weeks, on average
Progression-free Survival (PFS) | Up to 30 weeks, on average

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Yale University, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cance Center, New York, New York
  - Sarah Cannon Cancer Center, Nashville, Tennessee
- Institut Gustave Roussy, Villejuif, France
- Hospital Universitario Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Heist RS, Gounder MM, Postel-Vinay S, Wilson F, Garralda E, Do K, Shapiro GI, Martin-Romano P, Wulf G, Cooper M, Almon C, Nabhan S, Iyer V, Zhang Y, Marks K, Aguado-Fraile E, Basile F, Flaherty K, Burris HA. A phase 1 trial of AG-270 in patients with advanced solid tumors or lymphoma with homozygous MTAP deletion [abstract]. Mol Cancer Ther 2019;18(12 Suppl):Abstract nr PR03. doi:10.1158/1535-7163.TARG-19-PR03
- [Derived] Gounder M, Johnson M, Heist RS, Shapiro GI, Postel-Vinay S, Wilson FH, Garralda E, Wulf G, Almon C, Nabhan S, Aguado-Fraile E, He P, Romagnoli M, Hossain M, Narayanaswamy R, Sadou-Dubourgnoux A, Cooper M, Askoxylakis V, Burris HA, Tabernero J. MAT2A inhibitor AG-270/S095033 in patients with advanced malignancies: a phase I trial. Nat Commun. 2025 Jan 6;16(1):423. doi: 10.1038/s41467-024-55316-5. PMID 39762248
- [Derived] Konteatis Z, Travins J, Gross S, Marjon K, Barnett A, Mandley E, Nicolay B, Nagaraja R, Chen Y, Sun Y, Liu Z, Yu J, Ye Z, Jiang F, Wei W, Fang C, Gao Y, Kalev P, Hyer ML, DeLaBarre B, Jin L, Padyana AK, Dang L, Murtie J, Biller SA, Sui Z, Marks KM. Discovery of AG-270, a First-in-Class Oral MAT2A Inhibitor for the Treatment of Tumors with Homozygous MTAP Deletion. J Med Chem. 2021 Apr 22;64(8):4430-4449. doi: 10.1021/acs.jmedchem.0c01895. Epub 2021 Apr 8. PMID 33829783
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Lay summary — https://clinicaltrials.servier.com/trial/a-phase-1-study-of-ag-270-in-the-treatment-of-subjects-with-advanced-solid-tumors-or-lymphoma-with-homozygous-deletion-of-mtap/ — Study summary in lay language